CLINICAL TRIAL: NCT01747655
Title: A Post Marketing Observational Study of Activities of Daily Living in Advanced Parkinson's Disease Patients With Early Troublesome Motor Fluctuations and Treated With Duodopa - a Multi-country Study - MONOTREAT
Brief Title: A Post Marketing Observational Study of Activities of Daily Living in Advanced Parkinson's Disease Patients With Early Troublesome Motor Fluctuations and Treated With Duodopa - a Multi-country Study
Acronym: MONOTREAT
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-893
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
Keywords: Early Observational Advanced; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Duodopa: Participants given Duodopa gel administered with a portable pump directly into the proximal small intestine by a jejunal extension tube of the percutaneous endoscopic gastrostomy (PEG-J)
- Standard of Care: Participants that return to oral or transdermal anti-parkinson's disease medications

SUMMARY:
Patients with advanced Parkinson's Disease experience a range in the severity of their motor fluctuations. The rationale for this Post Marketing Observational Study is to demonstrate the benefits of Duodopa treatment on Parkinson's Disease patients entering the advanced stage of the disease whose motor fluctuations have become troublesome and complicate management with oral therapy. The aim of this post-marketing observational study is to assess the effect of Duodopa treatment on activities of daily living in advanced Parkinson's Disease participants characterised by either 2-4 hours of "off" time or 2 hours of non-troublesome or troublesome dyskinesia daily, supported by a Unified Parkinson's Disease Rating Scale Total Score in the best "on" state of at least 40 points at baseline.

DETAILED DESCRIPTION:
Data are recorded from visits most closely aligned with the planned periods of Visit 0 (V0): Baseline (After decision to use the temporary naso-duodenal tube (approximately 2-14 days) and after signature of the Patient Authorization/Informed Consent Form); Visit 1 (V1): At discharge from hospital; Visit 2 (V2): 3 months after discharge; Visit 3 (V3): 6 months after discharge; Visit 4 (V4): 12 months after discharge.

All participants have a temporary naso-duodenal tube used initially with the infusion pump to determine if the participant responds favorably to this method of treatment and to optimize the dose of Duodopa before permanent treatment is started.

Participants who choose a treatment other than Duodopa after the temporary naso-duodenal test phase are considered for the Standard of Care group. Participants who go on to select Apomorphine pump or Deep Brain Stimulation at any stage are not eligible to continue in this group or to continue in the observational period of study.

Participants who continue to with Duodopa treatment after the the temporary naso-duodenal test phase are the Duodopa group.

ELIGIBILITY:
Inclusion Criteria:

* Has advanced levodopa-responsive Parkinson's disease
* The decision to treat with Duodopa is made by the physician in accordance with the local label (Summary of Product Characteristics; product label) prior to any decision to approach the patient to participate in this study
* Parkinson's Disease (PD) medicinal treatment is unchanged for at least four weeks prior to baseline
* Takes oral medication four or more times daily
* Either has 2-4 hours of "off" time or 2 hours of non-troublesome or troublesome dyskinesia daily supported by a Unified Parkinson's Disease Rating Scale (UPDRS) Total Score in the best "on" state of at least 40 points at baseline; based on documented medical history

Exclusion Criteria:

* Use of Deep Brain Stimulation (DBS), Apomorphine pump or Duodopa treatment prior to baseline visit
* Severe dementia based on a Mini-Mental State Examination (MMSE) of < 24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital clinic
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koray Onuk, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Temporary Naso-jejunal Tube Period
Arm/Group | Duodopa | Standard of Care
Started | 64 (Main Analysis Set (MAS): participants with baseline and 1 further visit and ≥ 1 Duodopa treatment) | 0
Completed | 64 | 0
Not Completed | 0 | 0
Period: PEG-J Period (Duodopa Treatment)
Arm/Group | Duodopa | Standard of Care
Started | 58 (Dudopa MAS: Participants in the MAS that received Duodopa via PEG-J.) | 6 (Participants in the MAS that returned to SoC (no PEG-J introduced; did not meet selection criteria))
Completed | 44 | 6
Not Completed | 14 | 0
Not completed — Investigator Decision (Medical Event) | 5 | 0
Not completed — Patient Decision | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: PEG-J Period (Continued Treatment)
Arm/Group | Duodopa | Standard of Care
Started | 41 | 15 (SoC MAS: 6 SoC participants plus 9 participants who received Duodopa via PEG-J then returned to SoC)
Completed | 41 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects in the MAS
Arm/Group | Duodopa
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) II (Activities of Daily Living) Score: Mean Change From Baseline to 12 Months After Hospital Discharge
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to 13 questions, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability. UPDRS scores during "On" time (when PD symptoms are well controlled by the drug) are presented. Last observation carried forward (LOCF) was used for missing data.
Time Frame: Baseline (Week 0) and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 47 | 14
units on a scale | -2.1 (6.9) | 1.4 (5.1)

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) II (Activities of Daily Living) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to 13 questions, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability. UPDRS scores during "On" time (when PD symptoms are well controlled by the drug) are presented. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=47,7) | -4.4 (5.6) | 0.9 (6.0)
  Change from baseline to 6 months (n=44,6) | -3.4 (4.9) | -1.5 (2.3)
  Change from baseline to 12 months (n=41,6) | -1.8 (7.1) | 0.5 (5.3)

3. Secondary Outcome: Percentage of Participants Who Continued With Jejunal Extension Tube of the Percutaneous Endoscopic Gastrostomy (PEG-J) Treatment
Description: The percentage of participants who continued with PEG-J treatment after treatment via temporary naso-jejunal tube.
Time Frame: 14 days
Population: MAS population
Measure: Number; unit: percentage of participants
Arm/Group | Duodopa
Number analyzed (Participants) | 64
percentage of participants | 90.6

4. Secondary Outcome: Primary Reasons for Discontinuing Duodopa Treatment or for Discontinuing the Study
Description: The primary reasons for stopping treatment with Duodopa or for discontinuing the study.
Time Frame: 12 months
Population: Participants in the MAS who stopped treatment with Duodopa or discontinued from study.
Measure: Number; unit: participants
Arm/Group | Duodopa
Number analyzed (Participants) | 23
participants
  Patient decision | 9
  Investigator decision (due to medical event) | 8
  Investigator decision (other than medical event) | 2
  Does not feel has adequate support after discharge | 1
  Does not wish to carry the pump / device system | 1
  Does not wish to undergo the PEG-J procedure | 1
  Lost to follow-up | 1

5. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Item 32 (Duration) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: The UPDRS IV questionnaire consists of 4 individual items that assess the degree of dyskinesias (Item 32: duration; Item 33: disability; and Item 34: pain) and clinical fluctuations (Item 39: percentage of "off" times of the waking day). Individual UPDRS IV item scores range from 0 to 4. Higher scores indicate a higher complication of therapy. Observed values are presented for each visit as well as LOCF at 12 months after discharge. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=47,6) | -0.5 (1.1) | -0.5 (0.8)
  Change from baseline to 6 months after (n=44,6) | -0.6 (1.0) | -0.5 (1.0)
  Change from baseline to 12 months (n=41,6) | -0.4 (1.2) | -0.2 (1.2)
  Change from baseline to 12 months LOCF (n=47,14) | -0.5 (1.2) | -0.4 (0.9)

6. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Item 33 (Disability) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: as for outcome 5
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=47,6) | -0.9 (0.9) | -0.3 (0.5)
  Change from baseline to 6 months (n=44,6) | -0.9 (1.0) | -0.3 (0.5)
  Change from baseline to 12 months (n=41,6) | -0.5 (1.1) | -0.5 (1.4)
  Change from baseline to 12 months LOCF (n=47,14) | -0.9 (1.1) | -0.6 (1.1)

7. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Item 34 (Pain) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: as for outcome 5
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=47,6) | -0.3 (0.8) | 0.2 (0.4)
  Change from baseline to 6 months (n=43,6) | -0.3 (0.8) | -0.3 (0.8)
  Change from baseline to 12 months (n=41,6) | -0.3 (0.7) | 0.3 (0.8)
  Change from baseline to 12 months LOCF (n=47,14) | -0.3 (0.8) | 0.0 (0.9)

8. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) IV (Complications of Therapy) Item 39 (Clinical Fluctuations) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: as for outcome 5
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=47,6) | -0.9 (1.0) | -0.5 (1.5)
  Change from baseline to 6 months (n=44,6 | -0.9 (0.9) | -0.7 (0.5)
  Change from baseline to 12 months (n=41,6) | -0.8 (0.8) | -0.3 (1.0)
  Change from baseline to 12 months LOCF (n=47,14) | -0.8 (0.9) | -0.4 (1.1)

9. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) III (Motor Examination) Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: The UPDRS III questionnaire consists of 14 questions on motor examinations rated from 0 (absent/normal) to 4 (extreme impairment). Questions 20-26 are multi-part questions in that they are evaluated separately for multiple body parts (for example, for the left and right hand). Counting each of these assessments leads to a total of 27 answers. The UPDRS III score ranges from 0 to 108 with higher values indicating greater impairment and was calculated as the sum of the 27 answers provided to the 14 questions. Observed values are presented for each visit as well as LOCF at 12 months after discharge. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=51) | -12.9 (16.2) | -6.3 (11.9)
  Change from baseline to 6 months (n=49) | -8.9 (12.3) | -17.0 (22.6)
  Change from baseline to 12 months (n=46) | -8.7 (12.6) | 0.3 (16.5)
  Change from baseline to 12 months LOCF (n=61) | -8.9 (12.6) | -8.7 (21.2)

10. Secondary Outcome: Non-Motor Symptoms Assessment Scale for Parkinson's Disease (NMSS Rating Scale) Total Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: Non-motor symptoms assessed over the previous month were scored with respect to severity (0 = none, 1 = mild, 2 = moderate, 3 = severe) and with respect to frequency (1 = rarely, 2 = often, 3 = frequent, 4 = very frequent). The total NMSS score ranges from 0 to 360 with higher values indicating greater impairment and was calculated as the sum of all individual score values. Observed values are presented for each visit as well as LOCF at 12 months after discharge. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  Change from baseline to 3 months (n=44,5) | -39.5 (38.0) | -8.0 (14.6)
  Change from baseline to 6 months (n=40,5) | -33.7 (33.1) | -45.0 (64.5)
  Change from baseline to 12 months (n=38,6) | -33.9 (40.6) | -10.3 (15.2)
  Change from baseline to 12 months LOCF (n=40,10) | -32.5 (40.1) | -32.7 (45.9)

11. Secondary Outcome: Parkinson's Disease Quality of Life Questionnaire (PDQ-8) Summary Index Score: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: Participants were asked to state how often they had encountered certain problems over the past four weeks using the following rating scale: Never (0), occasionally (1), sometimes (2), often (3), always or cannot do at all (4). The PDQ-8 summary index was derived as the sum of the single items divided by 32. Scores range from 0 to 100. A higher summary index score indicates a higher impairment of quality of life. Observed values are presented for each visit as well as LOCF at 12 months after discharge. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0), at discharge from hospital, and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa | Standard of Care
Number analyzed (Participants) | 58 | 15
units on a scale
  3 months after discharge (n=46,6) | -15.7 (17.8) | -2.6 (6.4)
  6 months after discharge (n=43,6) | -15.4 (17.2) | -10.9 (20.3)
  12 months after discharge (n=41,6) | -12.3 (20.6) | -3.6 (7.5)
  12 months after discharge LOCF (n=42,10) | -12.1 (20.4) | -8.1 (16.2)

12. Secondary Outcome: Healthcare Resource Utilization (HCRU) Number of Office Visits: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: Participants were asked about their utilization of healthcare resources within the previous 3 months, including total number of office visits, total number of visits at home for Parkinson's disease, total number of emergency situations (overnight hospital stay, visit at emergency room, calls for immediate assistance [family/friend)], and calls to 911/emergency), received assistance at home (family/friend or paid caregiver), and falls. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Duodopa
Number analyzed (Participants) | 64
office visits
  Baseline (n=64) | 8.7 (9.8)
  Change from baseline to 3 months (n=53) | -3.0 (8.0)
  Change from baseline to 6 months (n=49) | -2.7 (9.8)
  Change from baseline to 12 months (n=47) | -2.1 (18.5)

13. Secondary Outcome: Healthcare Resource Utilization (HCRU) Number of Visits at Home: Mean Change From Baseline to 3, 6, and 12 Months After Hospital Discharge
Description: as for outcome 12
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Mean (Standard Deviation); unit: visits at home
Arm/Group | Duodopa
Number analyzed (Participants) | 64
visits at home
  Baseline (n=64) | 11.2 (31.4)
  Change from baseline to 3 months (n=53) | 0.8 (25.8)
  Change from baseline to 6 months (n=49) | -1.0 (21.5)
  Change from baseline to 12 months (n=47) | 4.0 (31.5)

14. Secondary Outcome: Healthcare Resource Utilization (HCRU) Emergency Situations: Percentage of Participants With Emergency Situations at 3, 6, and 12 Months After Hospital Discharge
Description: Participants were asked about their utilization of healthcare resources within the previous 3 months, including total number of office visits, total number of visits at home for Parkinson's disease, total number of emergency situations (overnight hospital stay, visit at emergency room, calls for immediate assistance [family/friend)], and calls to 911/emergency), received assistance at home (family/friend or paid caregiver), and falls. n=the number of participants with data at given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Number; unit: percentage of participants
Arm/Group | Duodopa
Number analyzed (Participants) | 64
percentage of participants
  Overnight hospital stay at Baseline (n=64) | 14.1
  Overnight hospital stay at 3 months (n=53) | 9.4
  Overnight hospital stay at 6 months (n=49) | 10.2
  Overnight hospital stay at 12 months (n=47) | 6.4
  Visit at emergency room at Baseline (n=64) | 10.9
  Visit at emergency room at 3 months (n=53) | 3.8
  Visit at emergency room at 6 months (n=49) | 14.3
  Visit at emergency room at 12 months (n=47) | 8.5
  Calls for immediate assistance at Baseline (n=64) | 25.0
  Calls for immediate assistance at 3 months (n=53) | 26.4
  Calls for immediate assistance at 6 months (n=49) | 6.1
  Calls for immediate assistance at 12 months (n=46) | 4.3
  911/Emergency at Baseline (n=64) | 4.7
  911/Emergency at 3 months (n=53) | 1.9
  911/Emergency at 6 months (n=49) | 4.1
  911/Emergency at 12 months (n=46) | 4.3

15. Secondary Outcome: Healthcare Resource Utilization (HCRU) Received Assistance at Home: Percentage of Participants Who Received Assistance at Home at 3, 6, and 12 Months After Hospital Discharge
Description: as for outcome 14
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Number; unit: percentage of participants
Arm/Group | Duodopa
Number analyzed (Participants) | 64
percentage of participants
  Family/friend at Baseline (n=64) | 59.4
  Family/friend at 3 months (n=53) | 49.1
  Family/friend at 6 months (n=49) | 44.9
  Family/friend at 12 months (n=47) | 46.8
  Paid caregiver at Baseline (n=64) | 10.9
  Paid caregiver at 3 months (n=53) | 24.5
  Paid caregiver at 6 months (n=49) | 24.5
  Paid caregiver at 12 months (n=47) | 25.5

16. Secondary Outcome: Healthcare Resource Utilization (HCRU) Falls: Percentage of Participants With Falls at 3, 6, and 12 Months After Hospital Discharge
Description: Participants were asked about their utilization of healthcare resources within the previous 3 months , including total number of office visits, total number of visits at home for Parkinson's disease, total number of emergency situations (overnight hospital stay, visit at emergency room, calls for immediate assistance [family/friend)], and calls to 911/emergency), received assistance at home (family/friend or paid caregiver), and falls. n=the number of participants with data at baseline and given time point.
Time Frame: Baseline (Week 0) and 3, 6, and 12 months after hospital discharge
Population: MAS population
Measure: Number; unit: percentage of participants
Arm/Group | Duodopa
Number analyzed (Participants) | 64
percentage of participants
  Baseline (n=64) | 35.9
  3 months (n=53) | 17.0
  6 months (n=49) | 24.5
  12 months (n=47) | 14.9

ADVERSE EVENTS:
Time Frame: All adverse events were collected from Baseline (Week 0) to 12 months after discharge (up to 13 months).
Groups:
- Duodopa: Participants given Duodopa gel administered with a portable pump directly into the proximal small intestine by a jejunal extension tube of the percutaneous endoscopic gastrostomy
Arm/Group | Duodopa
Serious Adverse Events (participants affected / at risk) | 14/64
Other Adverse Events (participants affected / at risk) | 10/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodopa (N=64)
CARDIAC FAILURE (Cardiac disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
MELAENA (Gastrointestinal disorders) | 1
GAIT DISTURBANCE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
PYREXIA (General disorders) | 1
SUDDEN DEATH (General disorders) | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
STOMA SITE INFECTION (Infections and infestations) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
FASCIITIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
BASILAR ARTERY THROMBOSIS (Nervous system disorders) | 1
COGNITIVE DISORDER (Nervous system disorders) | 1
DYSTONIA (Nervous system disorders) | 1
HYPOGLYCAEMIC COMA (Nervous system disorders) | 1
MOTOR DYSFUNCTION (Nervous system disorders) | 1
SPASMODIC DYSPHONIA (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 1
ABNORMAL DREAMS (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
DOPAMINE DYSREGULATION SYNDROME (Psychiatric disorders) | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 2
POLYURIA (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
HYPOTENSION (Vascular disorders) | 1
PALLOR (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodopa (N=64)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
CATHETER SITE HAEMATOMA (General disorders) | 1
DEVICE DISLOCATION (General disorders) | 1
CELLULITIS (Infections and infestations) | 1
STOMA SITE INFECTION (Infections and infestations) | 2
STOMA SITE DISCHARGE (Injury, poisoning and procedural complications) | 1
STOMA SITE GRANULOMA (Injury, poisoning and procedural complications) | 2
WEIGHT DECREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
READING DISORDER (Psychiatric disorders) | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1
THERAPY CESSATION (Surgical and medical procedures) | 3
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Results for the SoC group should be interpreted with care due to the small number of patients. Also, when comparing the SoC and Duodopa groups one should be aware that patients of the SoC group may have had Duodopa treatment before returning to SoC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.